CLINICAL TRIAL: NCT06299566
Title: Exploring Perceptions on the Proposed Cystic Fibrosis Screening Protocol Incorporating Next Generation Sequencing
Brief Title: Perceptions of the CF Screening Protocol Incorporating NGS
Status: Completed | Type: Observational
Sponsor: King's College London (Other)
Collaborators: University of Warwick (Other); Coventry University (Other); Barts & The London NHS Trust (Other); Cystic Fibrosis Trust (Other)
Responsible Party: Sponsor
Other Study IDs: CF NGS
Record Dates: First submitted 2024-02-20; First posted 2024-03-08 (Actual); Last update posted 2024-03-08 (Actual); Status verified 2024-03

CONDITIONS: Cystic Fibrosis
MeSH Terms: conditions — Cystic Fibrosis

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- People with experience of cystic fibrosis: Adults or children with experience of CF.
- Health professionals: Health professionals with experience of caring for people with experience of CF.

SUMMARY:
Newborn bloodspot screening (from now on referred to as screening) for cystic fibrosis (CF) became part of the national screening programme in 2007. Screening for CF is also well established internationally. The current process works well but has some disadvantages: carrier reporting - which is not the intention of CF screening in the UK (~200 pa); need for repeat samples which can be costly and contribute to parental worry (~300 pa.); mutation panels not fully reflecting the ethnic diversity of the birth population; identification of children designated as CF screen positive, inconclusive diagnosis (CFSPID) which can cause uncertainty (~20-30 pa).

A trial of NGS in one centre in the UK, for one year found that it was technically feasible at reasonable cost and with an acceptable turn around time. In addition, the trial determined that using NGS could mitigate against some of the disadvantages described above.

The purpose of this piece of work was to:

1. Gather, compare and analyse the views of a range of stakeholders on the proposed CF screening protocol incorporating NGS.
2. Use the outcomes to inform discussions and decisions by the fetal, maternal and child health (FMCH) group and UK National Screening Committee (NSC) about the proposed protocol
3. Consider what generalisable information on the views of stakeholders on newborn screening could be generated from this exercise to inform other FMCH and UK NSC discussions
4. Evaluate and learn from the exercise to inform future stakeholder engagement activities by the UK NSC and screening programmes.

ELIGIBILITY:
Inclusion Criteria:

1. Adults aged over 18 years of age who:

   (i) Were diagnosed with CF in childhood (ii) Were diagnosed with CF as adults (including those who would have been identified as CFSPID if NBS had been available and reporting it) (iii) Are carriers of CF (including parents/relatives of children/adults with CF and adults identified via other routes e.g. private testing)
2. Parents (aged over 18 years) of children identified through NBS who:

   (iv) Have CF (v) Are carriers of CF (vi) Have a CFSPID designation (vii) Have received a false positive NBS result for CF (viii) Have received a false negative NBS result for CF
3. Children aged over 10 years of age* who:

   (ix) Have CF (x) Have a CFSPID designation (xi) Are carriers of CF and have been informed of their carrier status

   *Ten years of age has been chosen for both pragmatic reasons and because this represents the age at which children will begin preparing for transition to adult services and therefore a period of increased independence and/or preparing for specialist review
4. Professionals involved in processing and/or communicating positive NBS results for CF to families or supporting families in health, community or education settings e.g. doctors, nurses, geneticists, genetic counsellors, midwives, social workers, dieticians, physiotherapists, teachers, university lecturers, charities.

Exclusion Criteria:

Exclusion criteria for those affected by CF:

1. Adults or children with non CF related co-morbidities that are likely to influence their perception of the proposed CF screening protocol incorporating NGS
2. Parents whose child has died prior to being approached to be involved in the study
3. Adults or children unable to understand the PIS and give informed consent/assent respectively
4. Adults or children whose recruitment is contraindicated on psychosocial or medical grounds (identified by their health visitor or specialist team).

Exclusion criteria for professionals:

Those not involved in processing, communicating positive NBS results for CF to families or supporting families in health, community or education settings.

Ages: 10 Years to 99 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: People with experience of CF, CFSPID or carrier status and health professionals with experience of caring for them.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Actual)
Dates: Start 2022-01-19 (Actual); Primary Completion 2023-02-28 (Actual); Study Completion 2023-02-28 (Actual)

PRIMARY OUTCOMES:
Focus groups/interviews/questionnaires exploring stakeholder views of the proposed CF screening protocol incorporating NGS. | February 2023
  Focus groups/interviews/questionnaires exploring stakeholder views, experiences and conceptualized harms/benefits in relation to the proposed CF screening protocol incorporating NGS

SECONDARY OUTCOMES:
Focus groups/interviews/questionnaires exploring stakeholder views on equivocal, carrier, false positives/negatives results, late onset/uncertain conditions | February 2023
  Focus groups/interviews/questionnaires exploring stakeholder views on equivocal, carrier, false positives/negatives results, late onset/uncertain conditions identified early in life (infertility, potential CF), missed CF diagnoses, as well as the way these outcomes are prioritised and ordered when considering NGS for CF NBS
Q sorts used to develop data and materials FMCH and UK NSC can use to engage stakeholders | February 2023
  Q sorts used to develop data and materials FMCH and UK NSC can use to engage stakeholders more widely with discussions about a) the proposed protocol, and b) wider use of genomic testing in NBS
Surveys to explore principles of engagement for stakeholders | February 2023
  Surveys to explore principles of engagement for this population, building on the 'golden rules' but with context specific guidance under each that can be used in future commissioning

CONTACTS AND LOCATIONS:
Locations (1):
- King's College London, London, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided
Data are available on request from the corresponding author. The data are not publicly available due to ethical constraints

REFERENCES:
- [Derived] Moody L, Clarke S, Compton M, Hughson-Gill R, Boardman F, Clark C, Holder P, Bonham JR, Chudleigh J. Development of an Online Scenario-Based Tool to Enable Research Participation and Public Engagement in Cystic Fibrosis Newborn Screening: Mixed Methods Study. J Particip Med. 2025 Mar 6;17:e59686. doi: 10.2196/59686. PMID 40053726